CLINICAL TRIAL: NCT06821893
Title: Vagus Auricular Stimulation for Tinnitus
Acronym: VAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor of Otolaryngology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202411118
Record Dates: First submitted 2025-02-04; First posted 2025-02-12 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Tinnitus
Keywords: Audiology; Otolaryngology; Mindfulness Based Stress Reduction (MBSR); auricular branch of vagus nerve; neuromodulation; transcutaneous stimulation
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: This pilot study is a randomized, double-blinded controlled trial of adult participants with chronic, moderate to severe bothersome subjective tinnitus.
Who Masked: Participant, Investigator
Masking Description: The participants, and research team will be unaware of whether device A or B corresponds to the stimulation or sham device during the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vibrational stimulation + MBSR (Experimental): Each participant will wear the Auricular stimulation device during the 30 minutes mindfulness exercise portion of the 2-hour MBSR group sessions. Additionally, they will wear the devices during the 20-minute at-home MBSR activities for the remaining six days of the week, totaling 120 minutes. The total expected duration of device usage per week will be 2.5 hours or 150 minutes.
  Mindfulness Based Stress Reduction: This is a standardized and structured training session that was originally developed by Jon Kabat-Zinn. Its primary objective is to assist participants in accepting their current condition and eliminating negative associations with it. All study participants will receive MBSR
  Interventions: Device: Vibrational stimulation
- Sham + MBSR (Sham Comparator): Each participant will wear the Sham device device during the 30 minutes mindfulness exercise portion of the 2-hour MBSR group sessions. Additionally, they will wear the devices during the 20-minute at-home MBSR activities for the remaining six days of the week, totaling 120 minutes. The total expected duration of device usage per week will be 2.5 hours or 150 minutes.
  Mindfulness Based Stress Reduction: This is a standardized and structured training session that was originally developed by Jon Kabat-Zinn. Its primary objective is to assist participants in accepting their current condition and eliminating negative associations with it. All study participants will receive MBSR
  Interventions: Device: Sham

INTERVENTIONS:
Device: Vibrational stimulation — The auricular stimulation device produces continuous vibrational stimulation directly to the conchae of the auricle. It is designed to stimulate the vagus nerve for neuromodulation to treat a variety of clinical indications. The system includes a pulse generator and an ear electrode device. Participants will use a vibration motor in a custom-created soft plastic clip for the left ear.
  Each participant will receive their own device by mail, which they will wear during the the 30 minutes mindfulness exercise portion of the 2-hour MBSR group sessions. Additionally, they will wear the devices during the 20-minute at-home MBSR activities for the remaining six days of the week, totaling 120 minutes. The total expected duration of device usage per week will be 2.5 hours or 150 minutes.
  Other Names: Auricular Stimulation
  Arms: Vibrational stimulation + MBSR
Device: Sham — The sham device looks and is used identically to the auricular stimulation device, but does not produce vibrational stimulation. There will be no difference in the usage directions of the sham device compared to the stimulation device.
  Each participant will receive their own device by mail, which they will wear during the 30 minutes mindfulness exercise portion of the 2-hour MBSR group sessions. Additionally, they will wear the devices during the 20-minute at-home MBSR activities for the remaining six days of the week, totaling 120 minutes. The total expected duration of device usage per week will be 2.5 hours or 150 minutes.
  Other Names: Sham device
  Arms: Sham + MBSR

SUMMARY:
This pilot study is a randomized, double-blinded controlled trial of adult participants with chronic, moderate to severe bothersome subjective tinnitus. Participants will be randomly assigned to either an active auricular stimulation device group or a sham-control group.Both groups will also undergo virtual Mindfulness-Based Stress Reduction(MBSR) over 8 weeks to promote tinnitus bother reduction, and general well-being. Outcome measures will be assessed at baseline, end of intervention, and at 1-month post-intervention.

DETAILED DESCRIPTION:
Adults experiencing moderate to severe tinnitus have significant impairment in their quality of life. While Cognitive Behavioral Therapy (CBT) is the most effective treatment for tinnitus, its accessibility is limited. Alternative treatment options such as masking pose significant risks and have varying success rates in achieving tinnitus cessation. Given these limitations and risks, there is a need to explore alternative treatment options for tinnitus that are both effective and easily accessible. Transcutaneous electrical stimulation of the vagus nerve has been explored as a treatment option for tinnitus using different study designs with varying response rate. In contrary, this pilot study will provide valuable insights and preliminary evidence for the effectiveness of transcutaneous stimulation of the auricular branch of the vagus nerve (TABVN-stim) utilizing a novel device that produces vibrational stimulation mimicking physiological sensory input to the ABVN. This research provides preliminary evidence for a potentially safe, non-invasive, and easily applicable treatment option for those suffering from chronic bothersome tinnitus, ultimately improving their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Ability to read, write, speak, and understand English
* Bothersome tinnitus with initial TSSF score greater than 40 on screening
* Available for the entire period of the study including one month follow-up after completion of 8-week intervention period
* Access to internet-connected device(s) such as phone, tablet, or laptop with a camera

Exclusion Criteria:

* Age>70
* Pregnant or planning to become pregnant during the study period
* Previous participation in an auricular stimulation trial
* Currently on active treatment for tinnitus
* Have cochlear implant or other device that impedes usage of auricular stimulation device
* Tinnitus related to ear surgery, Meniere's disease, ear infections, or other ear pathology
* Substance abuse
* Unstable psychiatric disorders
* Patient Health Questionnaire (PHQ-9) score greater than 9 History of brain surgery
* History of traumatic brain injury
* History of bradycardia or bradyarythmias

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-07-27 (Actual)

PRIMARY OUTCOMES:
Responder proportion | Week 9
  The responder proportion will be defined as number of participants with >12- point change in Tinnitus Severity Short Form [TSSF] score at the end of treatment compared to baseline, divided by the total number of participants in each group.
  TSSF score ranges from 0 (mild) to 100 (severe) The responder proportion will be compared between the active and sham group.

SECONDARY OUTCOMES:
Proportion of adequate device users | Week 9
  Feasibility of the auricular device will be assessed by recording the duration of device usage each week, summed over 8 weeks, and calculated as a percentage of the total expected usage which is 2.5 hours(per week) x 8 for each participant.
  Participants with >80% device usage will be defined as adequate device users.
  The proportion of adequate users will be compared between the stimulation and sham groups
Adverse events | Week 9, and 13
  The summary of reported adverse events after 8-weeks of the study period, and after 4 weeks post-intervention will be compared between stimulation and sham groups.
Proportion of participants reporting improvement on CGI-I | Week 9 and 13
  Participants will rate their perception of their response to tinnitus treatment using the CGI-I scale.
  The proportion of participants reporting improvement will be calculated as the number of participants with a CGI-I score ≤3 (defined as reporting improvement) divided by the total number of participants in each group.
  The proportion will be compared between the active and sham group after 8 weeks of intervention, and at 4 weeks post-intervention.
  Clinical Global Impression of Improvement Scale:
  The CGI-I scale is a self-reported measure widely used in previous studies and adapted from validated scales used in psychiatric studies.
  Participants will answer the question, "Overall, how do you rate your response to tinnitus treatment?"
  It offers 7 response options ranging from: 1-Very Much Improved, 2-Much Improved, 3-Minimally Improved, 4-No Change, 5-Minimally Worse, 6-Much Worse, to 7-Very Much Worse.
Change in CGI-S | Week 9, and 13
  The change in CGI-S score from baseline after 8 weeks of intervention and 4 weeks post intervention will be compared between the active and sham group.
  Clinical Global Impression of Severity (CGI-S) Scale:
  The CGI-S scale assesses the perceived severity problem level of tinnitus symptoms, with 5 response options ranging from 1-"Not bothered", 2-"Bothered a little, but not much", 3-"Bothered more than a little, but not a lot", 4-"Bothered a lot", to 5-"Extremely bothered.
  It poses the question, "Please indicate the overall amount of disturbance or "bother" that you experience in your life as a result of your tinnitus."
Responder proportion at 4weeks post-intervention follow up | Week 13
  Responder proportion will be defined as number of participants with >12- point change in Tinnitus Severity Short Form [TSSF] score at 4 weeks after the end of treatment compared to baseline divided by the total number of participants in each group.
  TSSF score ranges from 0 (mild) to 100 (severe) The responder proportion will be compared between the active and sham group.

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batts S, Stankovic KM. Tinnitus prevalence, associated characteristics, and related healthcare use in the United States: a population-level analysis. Lancet Reg Health Am. 2024 Jan 6;29:100659. doi: 10.1016/j.lana.2023.100659. eCollection 2024 Jan. PMID 38269207
- [Background] Tang D, Li H, Chen L. Advances in Understanding, Diagnosis, and Treatment of Tinnitus. Adv Exp Med Biol. 2019;1130:109-128. doi: 10.1007/978-981-13-6123-4_7. PMID 30915704
- [Background] Beukes EW, Andersson G, Allen PM, Manchaiah V, Baguley DM. Effectiveness of Guided Internet-Based Cognitive Behavioral Therapy vs Face-to-Face Clinical Care for Treatment of Tinnitus: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Dec 1;144(12):1126-1133. doi: 10.1001/jamaoto.2018.2238. PMID 30286238
- [Background] Miller L. Cognitive behavioral therapy for patients suffering with tinnitus distress. JAAPA. 2023 Sep 1;36(9):13-16. doi: 10.1097/01.JAA.0000947036.33633.84. PMID 37561667
- [Background] Butt MF, Albusoda A, Farmer AD, Aziz Q. The anatomical basis for transcutaneous auricular vagus nerve stimulation. J Anat. 2020 Apr;236(4):588-611. doi: 10.1111/joa.13122. Epub 2019 Nov 19. PMID 31742681
- [Background] Hilz MJ. Transcutaneous vagus nerve stimulation - A brief introduction and overview. Auton Neurosci. 2022 Dec;243:103038. doi: 10.1016/j.autneu.2022.103038. Epub 2022 Sep 27. PMID 36201901
- [Background] Kim AY, Marduy A, de Melo PS, Gianlorenco AC, Kim CK, Choi H, Song JJ, Fregni F. Safety of transcutaneous auricular vagus nerve stimulation (taVNS): a systematic review and meta-analysis. Sci Rep. 2022 Dec 21;12(1):22055. doi: 10.1038/s41598-022-25864-1. PMID 36543841
- [Background] Byun YJ, Lee JA, Nguyen SA, Rizk HG, Meyer TA, Lambert PR. Transcutaneous Electrical Nerve Stimulation for Treatment of Tinnitus: A Systematic Review and Meta-analysis. Otol Neurotol. 2020 Aug;41(7):e767-e775. doi: 10.1097/MAO.0000000000002712. PMID 32472915
- [Background] Meikle MB, Henry JA, Griest SE, Stewart BJ, Abrams HB, McArdle R, Myers PJ, Newman CW, Sandridge S, Turk DC, Folmer RL, Frederick EJ, House JW, Jacobson GP, Kinney SE, Martin WH, Nagler SM, Reich GE, Searchfield G, Sweetow R, Vernon JA. The tinnitus functional index: development of a new clinical measure for chronic, intrusive tinnitus. Ear Hear. 2012 Mar-Apr;33(2):153-76. doi: 10.1097/AUD.0b013e31822f67c0. PMID 22156949
- [Background] Langguth B, De Ridder D. Minimal Clinically Important Difference of Tinnitus Outcome Measurement Instruments-A Scoping Review. J Clin Med. 2023 Nov 15;12(22):7117. doi: 10.3390/jcm12227117. PMID 38002730
- [Background] Frumkin MR, Kallogjeri D, Piccirillo JF, Beukes EW, Manchaiah V, Andersson G, Rodebaugh TL. Development and Preliminary Evaluation of the Tinnitus Severity Short Form. Am J Audiol. 2021 Jun 14;30(2):404-415. doi: 10.1044/2021_AJA-20-00164. Epub 2021 May 24. PMID 34029120
- [Background] Natarajan N, Batts S, Stankovic KM. Noise-Induced Hearing Loss. J Clin Med. 2023 Mar 17;12(6):2347. doi: 10.3390/jcm12062347. PMID 36983347
- [Background] Kang HJ, Kang DW, Kim SS, Oh TI, Kim SH, Yeo SG. Analysis of Chronic Tinnitus in Noise-Induced Hearing Loss and Presbycusis. J Clin Med. 2021 Apr 19;10(8):1779. doi: 10.3390/jcm10081779. PMID 33921850
- [Background] Saeed S, Khan QU. The Pathological Mechanisms and Treatments of Tinnitus. Discoveries (Craiova). 2021 Sep 30;9(3):e137. doi: 10.15190/d.2021.16. eCollection 2021 Jul-Sep. PMID 35350720
- [Background] Dehaene S, Kerszberg M, Changeux JP. A neuronal model of a global workspace in effortful cognitive tasks. Proc Natl Acad Sci U S A. 1998 Nov 24;95(24):14529-34. doi: 10.1073/pnas.95.24.14529. PMID 9826734
- [Background] Hinkley LBN, Larson PS, Henderson Sabes J, Mizuiri D, Demopoulos C, Adams ME, Neylan TC, Hess CP, Nagarajan SS, Cheung SW. Striatal networks for tinnitus treatment targeting. Hum Brain Mapp. 2022 Feb 1;43(2):633-646. doi: 10.1002/hbm.25676. Epub 2021 Oct 5. PMID 34609038
- [Background] De Ridder D, Vanneste S, Congedo M. The distressed brain: a group blind source separation analysis on tinnitus. PLoS One. 2011;6(10):e24273. doi: 10.1371/journal.pone.0024273. Epub 2011 Oct 6. PMID 21998628
- [Background] Moller AR. Sensorineural Tinnitus: Its Pathology and Probable Therapies. Int J Otolaryngol. 2016;2016:2830157. doi: 10.1155/2016/2830157. Epub 2016 Feb 8. PMID 26977153
- [Background] Rademaker MM, Stegeman I, Ho-Kang-You KE, Stokroos RJ, Smit AL. The Effect of Mindfulness-Based Interventions on Tinnitus Distress. A Systematic Review. Front Neurol. 2019 Nov 1;10:1135. doi: 10.3389/fneur.2019.01135. eCollection 2019. PMID 31736854
- [Background] Noble W. Treatments for tinnitus. Trends Amplif. 2008 Sep;12(3):236-41. doi: 10.1177/1084713808320552. Epub 2008 Jul 17. PMID 18635586
- [Background] Garin P, Gilain C, Van Damme JP, de Fays K, Jamart J, Ossemann M, Vandermeeren Y. Short- and long-lasting tinnitus relief induced by transcranial direct current stimulation. J Neurol. 2011 Nov;258(11):1940-8. doi: 10.1007/s00415-011-6037-6. Epub 2011 Apr 21. PMID 21509429
- [Background] Lee HY. Adjunctive Role of Bifrontal Transcranial Direct Current Stimulation in Distressed Patients with Severe Tinnitus. J Korean Med Sci. 2019 Jan 4;34(3):e19. doi: 10.3346/jkms.2019.34.e19. eCollection 2019 Jan 21. PMID 30662385
- [Background] Cheung SW, Racine CA, Henderson-Sabes J, Demopoulos C, Molinaro AM, Heath S, Nagarajan SS, Bourne AL, Rietcheck JE, Wang SS, Larson PS. Phase I trial of caudate deep brain stimulation for treatment-resistant tinnitus. J Neurosurg. 2019 Sep 24;133(4):992-1001. doi: 10.3171/2019.4.JNS19347. Print 2020 Oct 1. PMID 31553940
- [Background] Hesser H, Weise C, Westin VZ, Andersson G. A systematic review and meta-analysis of randomized controlled trials of cognitive-behavioral therapy for tinnitus distress. Clin Psychol Rev. 2011 Jun;31(4):545-53. doi: 10.1016/j.cpr.2010.12.006. Epub 2010 Dec 23. PMID 21237544
- [Background] Fuller T, Cima R, Langguth B, Mazurek B, Vlaeyen JW, Hoare DJ. Cognitive behavioural therapy for tinnitus. Cochrane Database Syst Rev. 2020 Jan 8;1(1):CD012614. doi: 10.1002/14651858.CD012614.pub2. PMID 31912887
- [Background] Rodrigo H, Beukes EW, Andersson G, Manchaiah V. Internet-based cognitive-behavioural therapy for tinnitus: secondary analysis to examine predictors of outcomes. BMJ Open. 2021 Aug 20;11(8):e049384. doi: 10.1136/bmjopen-2021-049384. PMID 34417217
- [Background] Landry EC, Sandoval XCR, Simeone CN, Tidball G, Lea J, Westerberg BD. Systematic Review and Network Meta-analysis of Cognitive and/or Behavioral Therapies (CBT) for Tinnitus. Otol Neurotol. 2020 Feb;41(2):153-166. doi: 10.1097/MAO.0000000000002472. PMID 31743297
- [Background] Mueller L, Kallogjeri D, Frumkin MR, Dizdar K, Shin J, Rodebaugh T, Piccirillo JF. Predictors of Response to Cognitive Behavioral Therapy in Patients With Tinnitus. JAMA Otolaryngol Head Neck Surg. 2024 Sep 1;150(9):819-826. doi: 10.1001/jamaoto.2024.2264. PMID 39088223
- [Background] Kaldo V, Cars S, Rahnert M, Larsen HC, Andersson G. Use of a self-help book with weekly therapist contact to reduce tinnitus distress: a randomized controlled trial. J Psychosom Res. 2007 Aug;63(2):195-202. doi: 10.1016/j.jpsychores.2007.04.007. PMID 17662757
- [Background] Zenner HP, Vonthein R, Zenner B, Leuchtweis R, Plontke SK, Torka W, Pogge S, Birbaumer N. Standardized tinnitus-specific individual cognitive-behavioral therapy: a controlled outcome study with 286 tinnitus patients. Hear Res. 2013 Apr;298:117-25. doi: 10.1016/j.heares.2012.11.013. Epub 2012 Dec 31. PMID 23287811
- [Background] McKenna L, Marks EM, Hallsworth CA, Schaette R. Mindfulness-Based Cognitive Therapy as a Treatment for Chronic Tinnitus: A Randomized Controlled Trial. Psychother Psychosom. 2017;86(6):351-361. doi: 10.1159/000478267. Epub 2017 Nov 3. PMID 29131084
- [Background] McKenna L, Marks EM, Vogt F. Mindfulness-Based Cognitive Therapy for Chronic Tinnitus: Evaluation of Benefits in a Large Sample of Patients Attending a Tinnitus Clinic. Ear Hear. 2018 Mar/Apr;39(2):359-366. doi: 10.1097/AUD.0000000000000491. PMID 28945659
- [Background] Kreuzer PM, Goetz M, Holl M, Schecklmann M, Landgrebe M, Staudinger S, Langguth B. Mindfulness-and body-psychotherapy-based group treatment of chronic tinnitus: a randomized controlled pilot study. BMC Complement Altern Med. 2012 Nov 28;12:235. doi: 10.1186/1472-6882-12-235. PMID 23186556
- [Background] Vernon JA, Meikle MB. Masking devices and alprazolam treatment for tinnitus. Otolaryngol Clin North Am. 2003 Apr;36(2):307-20, vii. doi: 10.1016/s0030-6665(02)00163-9. PMID 12856299
- [Background] Bahmad F Jr, Carasek N, Lamounier P. Cochlear implant in tinnitus management. Curr Opin Otolaryngol Head Neck Surg. 2023 Apr 1;31(2):155-157. doi: 10.1097/MOO.0000000000000874. Epub 2023 Jan 31. PMID 36912228
- [Background] Rufener KS, Wienke C, Salanje A, Haghikia A, Zaehle T. Effects of transcutaneous auricular vagus nerve stimulation paired with tones on electrophysiological markers of auditory perception. Brain Stimul. 2023 Jul-Aug;16(4):982-989. doi: 10.1016/j.brs.2023.06.006. Epub 2023 Jun 17. PMID 37336282
- [Background] Vanneste S, Plazier M, Van de Heyning P, De Ridder D. Transcutaneous electrical nerve stimulation (TENS) of upper cervical nerve (C2) for the treatment of somatic tinnitus. Exp Brain Res. 2010 Jul;204(2):283-7. doi: 10.1007/s00221-010-2304-5. Epub 2010 May 28. PMID 20505927
- [Background] Botha C, Farmer AD, Nilsson M, Brock C, Gavrila AD, Drewes AM, Knowles CH, Aziz Q. Preliminary report: modulation of parasympathetic nervous system tone influences oesophageal pain hypersensitivity. Gut. 2015 Apr;64(4):611-7. doi: 10.1136/gutjnl-2013-306698. Epub 2014 May 28. PMID 24870622
- [Background] Cutsforth-Gregory JK, Benarroch EE. Nucleus of the solitary tract, medullary reflexes, and clinical implications. Neurology. 2017 Mar 21;88(12):1187-1196. doi: 10.1212/WNL.0000000000003751. Epub 2017 Feb 15. No abstract available. PMID 28202704
- [Background] Steenerson RL, Cronin GW. Tinnitus reduction using transcutaneous electrical stimulation. Otolaryngol Clin North Am. 2003 Apr;36(2):337-44. doi: 10.1016/s0030-6665(02)00164-0. PMID 12856301
- [Background] Yakunina N, Kim SS, Nam EC. BOLD fMRI effects of transcutaneous vagus nerve stimulation in patients with chronic tinnitus. PLoS One. 2018 Nov 28;13(11):e0207281. doi: 10.1371/journal.pone.0207281. eCollection 2018. PMID 30485375
- [Background] Yap JYY, Keatch C, Lambert E, Woods W, Stoddart PR, Kameneva T. Critical Review of Transcutaneous Vagus Nerve Stimulation: Challenges for Translation to Clinical Practice. Front Neurosci. 2020 Apr 28;14:284. doi: 10.3389/fnins.2020.00284. eCollection 2020. PMID 32410932
- [Background] Qureshi IS, Datta-Chaudhuri T, Tracey KJ, Pavlov VA, Chen ACH. Auricular neural stimulation as a new non-invasive treatment for opioid detoxification. Bioelectron Med. 2020 Mar 30;6:7. doi: 10.1186/s42234-020-00044-6. eCollection 2020. PMID 32266304
- [Background] Lee SK, Chung H, Chung JH, Yeo SG, Park MS, Byun JY. Effectiveness of transcutaneous electrical stimulation for chronic tinnitus. Acta Otolaryngol. 2014 Feb;134(2):159-67. doi: 10.3109/00016489.2013.844854. Epub 2013 Nov 11. PMID 24215217
- [Background] Engelberg M, Bauer W. Transcutaneous electrical stimulation for tinnitus. Laryngoscope. 1985 Oct;95(10):1167-73. doi: 10.1288/00005537-198510000-00003. PMID 3900611
- [Background] Aydemir G, Tezer MS, Borman P, Bodur H, Unal A. Treatment of tinnitus with transcutaneous electrical nerve stimulation improves patients' quality of life. J Laryngol Otol. 2006 Jun;120(6):442-5. doi: 10.1017/S0022215106000910. Epub 2006 Mar 24. PMID 16556347
- [Background] Tan G, Adams J, Donovan K, Demarest P, Willie JT, Brunner P, Gorlewicz JL, Leuthardt EC. Does vibrotactile stimulation of the auricular vagus nerve enhance working memory? A behavioral and physiological investigation. Brain Stimul. 2024 Mar-Apr;17(2):460-468. doi: 10.1016/j.brs.2024.04.002. Epub 2024 Apr 7. PMID 38593972
- [Background] Addorisio ME, Imperato GH, de Vos AF, Forti S, Goldstein RS, Pavlov VA, van der Poll T, Yang H, Diamond B, Tracey KJ, Chavan SS. Investigational treatment of rheumatoid arthritis with a vibrotactile device applied to the external ear. Bioelectron Med. 2019 Apr 17;5:4. doi: 10.1186/s42234-019-0020-4. eCollection 2019. PMID 32232095
- [Background] Gos E, Rajchel JJ, Dziendziel B, Kutyba J, Bienkowska K, Swierniak W, Gocel M, Raj-Koziak D, Skarzynski PH, Skarzynski H. How to Interpret Tinnitus Functional Index Scores: A Proposal for a Grading System Based on a Large Sample of Tinnitus Patients. Ear Hear. 2021 May/Jun;42(3):654-661. doi: 10.1097/AUD.0000000000000967. PMID 33156124
- [Background] Gos E, Sagan A, Skarzynski PH, Skarzynski H. Improved measurement of tinnitus severity: Study of the dimensionality and reliability of the Tinnitus Handicap Inventory. PLoS One. 2020 Aug 25;15(8):e0237778. doi: 10.1371/journal.pone.0237778. eCollection 2020. PMID 32841249
- [Background] Henry JA, Griest S, Thielman E, McMillan G, Kaelin C, Carlson KF. Tinnitus Functional Index: Development, validation, outcomes research, and clinical application. Hear Res. 2016 Apr;334:58-64. doi: 10.1016/j.heares.2015.06.004. Epub 2015 Jun 12. PMID 26074306
- [Background] Kallogjeri D, Spitznagel EL Jr, Piccirillo JF. Importance of Defining and Interpreting a Clinically Meaningful Difference in Clinical Research. JAMA Otolaryngol Head Neck Surg. 2020 Feb 1;146(2):101-102. doi: 10.1001/jamaoto.2019.3744. No abstract available. PMID 31804662
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Polak T, Markulin F, Ehlis AC, Langer JB, Ringel TM, Fallgatter AJ. Far field potentials from brain stem after transcutaneous vagus nerve stimulation: optimization of stimulation and recording parameters. J Neural Transm (Vienna). 2009 Oct;116(10):1237-42. doi: 10.1007/s00702-009-0282-1. PMID 19728032
- [Background] Santorelli, S., Mindfulness-based stress reduction (MBSR): Standards of practice. 2014: Center for Mindfulness in Medicine, Health Care & Society, University of Massachusetts Medical School, 2014